CLINICAL TRIAL: NCT00246714
Title: Pathophysiology and Clinical Relevance of Endotoxin Tolerance in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: P.Pickkers, Radboud University Medical Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PP03
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Endotoxemia
Keywords: endotoxin tolerance; humans; cross-tolerance; pro and anti-inflammatory cytokines
MeSH Terms: conditions — Endotoxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repeated injections of endotoxin during 5 days

SUMMARY:
A number of diseases lead to a so called systemic inflammatory response syndrome (SIRS). This excessive response is self-destructive and leads to major complications of the initial disease: dysfunction of the microcirculation, systemic vasodilation, and increased capillary leakage and oedema. Animal studies have shown that pre-treatment with endotoxin (lipopolysaccharide or LPS) suppress the excessive immune response and when rechallenged, the animal survive a normally lethal dose of endotoxin.

Besides a diminished cytokine response, an increased production of leucocytes in the bone marrow and an increased phagocytosis after pre-treatment with endotoxin is seen. The combination of these factors: diminished systemic inflammatory response and increased cellular immunity makes that endotoxin tolerance is a useful tool for preventing the complications after an excessive inflammatory response.

Further, the presence of cross-tolerance has also been shown: Endotoxin tolerant mice survive more after induction of a normally lethal fungal infection. Endotoxin tolerance is also protective for ischemia/reperfusion injury in kidneys, heart and liver. Little data is known about endotoxin tolerance in human.

The purpose of this study is to induce a state of tolerance through 2 different administration schedules and monitor the effect of tolerance on pro- and anti-inflammatory cytokines, other inflammatory parameters and different proteins involved in the signalling pathway. The effects of tolerance on vascular reactivity will be determined. Finally, the effect of tolerance on ischemia-reperfusion injury will be investigated.

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* drug-, nicotine-, alcohol abuses
* tendency towards fainting
* BMI < 18 kg/m2

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
inducing endotoxin tolerance | 5 days
Hemodynamics | 5 days
Markers of Inflammation | 5 days
Cytokines | 5 days
Mediators of Vascular reactivity | 5 days
Sensitivity to norepinephrine | 5 days
Endothelial-dependent vasorelaxation | 5 days
Cross tolerance | 6 days
Ischemia-reperfusion injury | 6 days
Effects on tissue saturation (measured by NIRS) | 24 hrs after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands